CLINICAL TRIAL: NCT06717425
Title: A PHASE 2A, RANDOMIZED, DOUBLE-BLIND, SPONSOR-OPEN, PLACEBO-CONTROLLED, PARALLEL GROUP, DOSE-RANGING STUDY OF PF-07976016 TO ASSESS SAFETY AND EFFICACY IN ADULT PARTICIPANTS WITH OBESITY
Brief Title: A Study to Learn About the Study Medicine Called PF-07976016 in Adults With Obesity
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C5541010; 2024-513679-42-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2024-12-02; First posted 2024-12-05 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Obesity
Keywords: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: This is a randomized, double-blind (investigator and participant), sponsor-open, placebo-controlled study.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- PF-07976016 Dose 1 (Experimental)
  Interventions: Drug: PF-07976016
- PF-07976016 Dose 2 (Experimental)
  Interventions: Drug: PF-07976016
- PF-07976016 Dose 3 (Experimental)
  Interventions: Drug: PF-07976016
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PF-07976016 — Taken once daily
  Arms: PF-07976016 Dose 1; PF-07976016 Dose 2; PF-07976016 Dose 3
Drug: Placebo — Taken once daily
  Arms: Placebo

SUMMARY:
The purpose of this clinical trial is to learn about the safety and effects of the study medicine (called PF-07976016) for the potential treatment of obesity. The study will compare the experiences of participants taking the study medicine (PF-07976016) to those of participants who take placebo (a lookalike substance that contains no active study medicine). The aim is to measure the body's response to the study medicine, including any changes in participants' body weight and how well they tolerate the study medicine.

ELIGIBILITY:
Key Inclusion Criteria:

* Male or non-pregnant, non-breastfeeding female, 18 to 74 years of age at Visit 1
* Body Mass Index ≥30.0 kg/m2 at Visit 1, with stable body weight, defined as <5 kg change in the 12 weeks before Visit 1
* Eligible and willing to receive required background medicine
* Willing and able to comply with all study procedures

Key Exclusion Criteria:

* Any medical or psychiatric condition or laboratory abnormality, or recent serious illness or hospitalization, that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study including diagnosis of type 2 diabetes mellitus, type 1 or secondary forms of diabetes.
* Use of any prohibited prior or concomitant medication(s)
* Presence of specified abnormalities on diagnostic assessments including clinical laboratory tests at Visit 1.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 263 (Actual)
Dates: Start 2024-12-09 (Actual); Primary Completion 2025-10-23 (Actual); Study Completion 2026-01-12 (Actual)

PRIMARY OUTCOMES:
Percent change from baseline in body weight | Baseline to Week 16

SECONDARY OUTCOMES:
Number of participants with treatment emergent adverse events | From first dose (Day 1) up to 28-35 days after final dose, a total of approximately 21 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (37):
- United States (27):
  - Anaheim Clinical Trials, LLC, Anaheim, California
  - Artemis Institute for Clinical Research, San Diego, California
  - Clinical & Translational Research Center, Aurora, Colorado
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - Westside Center for Clinical Research, Jacksonville, Florida
  - New Horizon Research Center, Miami, Florida
  - Renstar Medical Research, Ocala, Florida
  - St Johns Center for Clinical Research, Saint Augustine, Florida
  - Rophe Adult and Pediatric Medicine/SKYCRNG, Union City, Georgia
  - East-West Medical Research Institute, Honolulu, Hawaii
  - Cotton O'Neil Diabetes & Endocrinology, Topeka, Kansas
  - L-MARC Research Center, Louisville, Kentucky
  - Pennington Biomedical Research Center, Baton Rouge, Louisiana
  - StudyMetrix Research, City of Saint Peters, Missouri
  - Rochester Clinical Research, LLC, Rochester, New York
  - Accellacare - Wilmington, Wilmington, North Carolina
  - AMR Clinical, Norman, Oklahoma
  - Cornerstone Nutrition and Diabetes, Norman, Oklahoma
  - Capital Area Research, LLC, Camp Hill, Pennsylvania
  - Elligo Clinical Research Center, Austin, Texas
  - Texas Diabetes & Endocrinology, P.A., Austin, Texas
  - Velocity Clinical Research, Dallas, Dallas, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - Consano Clinical Research, LLC, Shavano Park, Texas
  - Chrysalis Clinical Research, St. George, Utah
  - Southwest Internal Medicine, PC, St. George, Utah
  - Selma Medical Associates, Winchester, Virginia
- Canada (5):
  - Ocean West Research Clinic, Surrey, British Columbia
  - Dawson Clinical Research Inc., Guelph, Ontario
  - The Wharton Medical Clinic Clinical Trials Inc., Hamilton, Ontario
  - Milestone Research Inc., London, Ontario
  - Canadian Phase Onward, Toronto, Ontario
- Poland (5):
  - Centrum Zdrowia Metabolicznego Pawel Bogdanski, Poznan, Greater Poland Voivodeship
  - Medicome Sp. z o. o., Oświęcim, Lesser Poland Voivodeship
  - Ekamed, Lublin, Lublin Voivodeship
  - Centrum Badan Klinicznych PI-House sp. z o.o., Gdansk, Pomeranian Voivodeship
  - Centrum Medyczne Pratia Gdynia, Gdynia, Pomeranian Voivodeship

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C5541010